CLINICAL TRIAL: NCT07397728
Title: TREX1 Gene Mutations and Their Role in Systemic Lupus Erythematosus: A Genotype-Phenotype Correlation Study
Brief Title: " TREX1 Gene Mutations and Their Role in Systemic Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Amira Rabea AbuElfadl, Resident at Dermatology , venereology and andrology, Faculty of medicine, South Valley University
Other Study IDs: TREX1 Gene
Record Dates: First submitted 2026-01-23; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample Collection: DNA extracted from 4 mL EDTA blood from SLE patients and healthy controls.
  Genotyping: Real-time polymerase chain reaction (PCR) genotyping for TREX1 will be done with the TaqMan-Allelic discrimination method in a Step One Plus Real-Time PCR system (Applied Biosystems, Foster City, CA, USA), and the results will be analyzed using the Allelic Discrimination software program (Applied Biosystems).
  Mutation Analysis: Variants will be compared to reference sequences (e.g., NM_016381.3) and classified according to ACMG guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A : (Systemic Lupus Erythrematosus): About 60 patients ) diagnosed with SLE based on 2019 EULAR/ACR criteria, each with at least one cutaneous manifestation.
  Interventions: Diagnostic Test: TREX1 gene polymorphisms
- Group B (Healthy Controls): 30 age- and sex-matched healthy controls with no personal or family history of autoimmune disease and negative ANA and anti-dsDNA.
  Interventions: Diagnostic Test: TREX1 gene polymorphisms

INTERVENTIONS:
Diagnostic Test: TREX1 gene polymorphisms — To assess the prevalence of selected autoantibodies as (anti-dsDNA, anti-Sm, anti-Ro/SSA, anti-La/SSB) and TREX1 gene polymorphisms in SLE patients, and their association with clinical features and disease activity
  Other Names: anti-dsDNA, anti-Sm, anti-Ro/SSA, anti-La/SSB

SUMMARY:
Systemic lupus erythematosus (SLE) is a multisystem autoimmune disease characterized by diverse clinical manifestations, prominently involving the skin.

DETAILED DESCRIPTION:
Cutaneous lesions are among the earliest and most frequent features of SLE, with over 70% of patients developing mucocutaneous involvement during their disease course.

The presence and severity of cutaneous manifestations have been associated with specific autoantibodies, such as anti-Ro/SSA and anti-dsDNA, which may reflect underlying genetic susceptibility.

Recent studies have also implicated gene polymorphisms in IRF5, STAT4, TREX1, and TNFA in the pathogenesis of cutaneous SLE phenotypes.

Defective TREX1 exonuclease activity, leading to intracellular accumulation of DNA, may trigger type I interferon activation-a key mechanism in lupus pathophysiology.

Despite the extensive global literature, data from Egyptian patients remain limited, especially regarding the relationship between TREX1 gene variants and cutaneous lupus phenotypes.

Understanding how autoantibody profiles and gene polymorphisms relate to clinical features and disease activity could enhance early diagnosis, predict flares, and improve personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-60 years
* Diagnosed as SLE per 2019 EULAR/ACR classification criteria.
* Presence of at least one cutaneous manifestation (acute, subacute, or chronic).
* Willing to provide written informed consent for participation and genetic testing

Exclusion Criteria:

* Overlap autoimmune syndromes (e.g., dermatomyositis, systemic sclerosis).
* Systemic infection, malignancy, or pregnancy.
* Use of biologic therapy or immunosuppressive pulses within one month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Group A: 60 adults (18-60 years) diagnosed with SLE based on 2019 EULAR/ACR criteria, each with at least one cutaneous manifestation.
  * Group B: 30 age- and sex-matched healthy controls with no personal or family history of autoimmune disease and negative ANA and anti-dsDNA.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus Assessment | 3 Months
  Assessment of disease activity in Systemic Lupus Erythematosus (SLE) using Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K). SLEDAI-2K as follows :
  1-5 is Mild disease activity 6-10 is Moderate disease activity 11 or more is Severe disease activity
TREX1 gene polymorphism and SLE | 3 Months
  Assessment the association between TREX1 gene polymorphism and systemic lupus erythematosus susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Mohammed Hegazy, Professor, Study Chair — Dermatology, Venereology and Andrology. Faculty of Medicine,Qena University; Mohammed Hosny Hassan, Professor, Study Director — Biochemistry ,Qena faculty of medicine ,south valley university
Locations (1):
- Qina University hospital, South Valley University Hospital, Qina, South Valley, Egypt

IPD SHARING:
Plan to Share IPD: Undecided